CLINICAL TRIAL: NCT03875495
Title: A Phase I/II Dose Escalation Study Evaluating Safety and Activity of Autologous CD34+-Enriched Hematopoietic Progenitor Cells Genetically Modified With a Lentiviral Vector Encoding for the Human Interferon-ɑ2 Gene in Multiple Myeloma Patients With Early Relapse After Intensive Front Line Therapy
Brief Title: A Phase I/II Study Evaluating Temferon in Multiple Myeloma Patients With Early Relapse After Front Line Therapy (TEM-MM)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Failure to recruit patients
Sponsor: Genenta Science (Industry)
Collaborators: IRCCS San Raffaele (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEM-MM-101
Record Dates: First submitted 2019-03-13; First posted 2019-03-14 (Actual); Results first posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Multiple Myeloma
Keywords: Temferon; Gene Therapy; Immunotherapy; Hematological malignancy
MeSH Terms: conditions — Multiple Myeloma; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temferon (Experimental): Autologous CD34+-enriched hematopoietic progenitor cells exposed ex vivo to a specific lentiviral vector encoding for the human IFN-ɑ2 gene.
  Its expression is tightly controlled by the human TIE2 enhancer/promoter sequence and by a post-transcriptional regulation layer represented by target miRNA sequences. This enables suppression of IFN-ɑ2 expression in HSPCs, thereby further increasing the specificity of the delivery strategy for their Tie2 expressing myeloid cell progeny.
  Interventions: Drug: Temferon

INTERVENTIONS:
Drug: Temferon — Genetically modified autologous HSPCs

SUMMARY:
This is a non-randomized, open label, phase I/II, dose-escalation study, involving a single injection of Temferon, an investigational advanced therapy consisting of autologous CD34+-enriched hematopoietic stem and progenitor cells exposed to transduction with a lentiviral vector driving myeloid-specific interferon-ɑ2 expression, which will be administered to up to 9 patients affected by multiple myeloma in early relapse after intensive front line treatment.

DETAILED DESCRIPTION:
This is a non-randomized, open label, single center, phase I/II, therapeutic exploratory, dose-escalation, prospective study, involving a single intravenous infusion of Temferon, an investigational advanced therapy consisting of autologous CD34+-enriched hematopoietic stem and progenitor cells (HSPCs) exposed to transduction with a third-generation, vesicular stomatitis virus-G (VSV-G) pseudo-typed lentiviral vector driving myeloid-specific interferon-ɑ2 (IFN-ɑ2) expression, which will be administered to up to 9 patients affected by multiple myeloma in early relapse after intensive front line treatment. The study will recruit, treat and follow-up patients at a specialist hematology and bone marrow transplantation unit at Ospedale San Raffaele (OSR) in Milan, Italy.

The study will enrol multiple myeloma patients that have experienced an early relapse after intensive front line treatment, have been treated with an approved second line combination treatment regimen and obtained at least a very good partial remission (VGPR) according to International Myeloma Working Group (IMWG) criteria. Once the written informed consent is obtained, and screening procedures have been completed, harvesting of HSPCs will occur. Patients will be offered maintenance treatment during Temferon production and release. Upon Temferon release for clinical use, patients will be admitted to the transplantation unit for receipt of a reduced-intensity conditioning regimen consisting of melphalan. This will be followed by autologous stem cell transplant (ASCT) and administration of Temferon. In-patient monitoring will occur until hematological recovery occurs. Thereafter, regular follow-up of patients will occur up to 2 years (+730 days). At the +730 day visit, patients will be invited to participate in a long term follow-up study which will last for an additional 6 years.

3 cohorts of 3 patients will receive escalating doses of Temferon.

In the event that MM disease progression occurs, patients will be managed according to best clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma patients with early relapse after intensive front-line treatment and disease measurable by serum biomarkers, who have obtained at least a VGPR after second-line salvage treatment.
* Able and willing to provide written informed consent.
* Able to comply with study protocol and procedures.
* Performance status scores: Eastern Cooperative Oncology Group (ECOG) < 2 and Karnofsky > 70%.
* Life expectancy of ≥ 6 months.
* Adequate cardiac, renal, hepatic and pulmonary functions as evidenced by (at screening and prior to conditioning):

  * Left ventricular ejection fraction (LVEF) ≥ 45% by echo and normal electrocardiogram (ECG) or presence of abnormalities not significant for cardiac disease. Absence of severe pulmonary hypertension;
  * Diffusing capacity of the lung for carbon monoxide (DLCO) >50% and forced expiratory volume in 1 sec (FEV1) and forced expiratory vital capacity (FVC) > 60% predicted (if non cooperative: pulse oximetry > 95 % in room air);
  * Serum creatinine < 2x ULN and estimated glomerular filtration rate (eGFR) > 30 ml/min/1.73m2;
  * Alkaline phosphatase (ALP), alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 2.5 x ULN, and total bilirubin ≤ 2.0 mg/dl.
* Women of child-bearing potential enrolled in the study must have a negative pregnancy test at screening and agree to use two distinct acceptable methods of contraception during the trial.
* Men enrolled in the study with partners who are women of child bearing potential, must be willing to use an acceptable barrier contraceptive method during the trial or have undergone successful vasectomy at least 6 months prior to entry into the study. Successful vasectomy needs to have been confirmed by semen analysis.

Exclusion Criteria:

* Use of other investigational agents within 4 weeks prior to experimental treatment (within 6 weeks if use of long-acting agents).
* Severe active viral, bacterial, or fungal infection at eligibility evaluation.
* Active autoimmune disease or a clinically relevant autoimmune manifestations, requiring immunosuppressive treatment, i.e. psoriasis, systemic lupus erythematosus, rheumatoid arthritis, vasculitis, immune-mediated peripheral neuropathies.
* Active sarcoidosis requiring steroid or other immunosuppressive treatment.
* Primary amyloidosis.
* History of neuropsychiatric illness including severe depression, schizophrenia, bipolar disorders, impaired cognitive function, dementia or suicidal tendency.
* Neuropathy > grade 2.
* History of severe cardiovascular disease such as prior stroke, coronary artery disease requiring intervention, unresolved arrhythmias.
* Malignant neoplasia (except local skin cancer or cervical intraepithelial neoplasia) or family history of familial cancer syndromes.
* Myelodysplasia, cytogenetic or molecular alterations specifically associated with clonal hematopoiesis of the myeloid lineage, or other serious hematological disorder other than the plasma cell dyscrasia.
* Other clinical conditions judged by the Investigator non-compatible with the study procedures.
* Positivity for HIV-1 or HIV-2 (serology or RNA), and/or Hepatitis B Virus Surface Antigen (HbsAg) and/or Hepatitis B Virus (HBV) DNA and/or Hepatitis C Virus (HCV) RNA (or negative HCV RNA but on antiviral treatment) and/or Treponema Pallidum or Mycoplasma active infection.
* Active alcohol or substance abuse within 6 months of the study.
* Pregnancy or lactation.
* Previous allogeneic bone marrow transplantation, kidney or liver transplant, or gene therapy.
* Prior to conditioning: inability to meet the target mobilization cell number needed to manufacture the Drug Product after at least 2 attempts of HSPC collection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Ciceri, MD, Principal Investigator — Ospedale San Raffaele, Milan, Italy
Locations (1):
- Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 patients recruited but none received Temferon. Unable to recruit additional patients due to the ongoing COVID-19 pandemic.
Groups:
- Temferon: Autologous CD34+-enriched hematopoietic progenitor cells exposed ex vivo to a specific lentiviral vector encoding for the human IFN-ɑ2 gene.
  Its expression is tightly controlled by the human TIE2 enhancer/promoter sequence and by a post-transcriptional regulation layer represented by target miRNA sequences. This enables suppression of IFN-ɑ2 expression in HSPCs, thereby further increasing the specificity of the delivery strategy for their Tie2 expressing myeloid cell progeny.
  Temferon: Genetically modified autologous HSPCs
Period: Overall Study
Arm/Group | Temferon
Started | 3
Completed | 0
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: No patients completed the baseline visit
Groups:
- Patient Recruitment: 3 patients recruited into the study but no patients received Temferon. Study terminated due to inability to recruit additional patients in view of the ongoing COVID-19 pandemic
Arm/Group | Patient Recruitment
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Race/Ethnicity, Customized
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Tolerability and Safety of Temferon Over the First 90 Days Following Administration as Determined by the Incidence of CTCAEs
Description: 0 participants analyzed. All the patients were withdrawn before treatment
Time Frame: 90 days
Population: Untreated patients
Groups:
- Untreated Patients: 3 Patients were recruited but did not receive Temferon
Arm/Group | Untreated Patients
Number analyzed (Participants) | 0

2. Secondary Outcome: Long Term Tolerability and Safety of Temferon as Determined by the Incidence of CTCAEs
Description: 0 participants analyzed. All the patients were withdrawn before treatment
Time Frame: 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Proportion of Patients Achieving Hematologic Recovery by Day +30 (Defined as the First of at Least 3 Consecutive Days With a Neutrophil Count >0.5 x 10^9/L and Platelet Count >20 x 10^9/L) in the Absence of Transfusions
Time Frame: 30 days
Reporting Status: Not Posted

4. Secondary Outcome: Determine the Maximum Tolerated Dose of Temferon
Time Frame: 30 days
Reporting Status: Not Posted

5. Secondary Outcome: Identify Presence of Transduced Myeloid Cells in Bone Marrow as Determined by Vector Copy Number
Time Frame: Up to 2 years
Reporting Status: Not Posted

6. Secondary Outcome: Identify Presence of Transduced Myeloid Cells in Peripheral Blood as Determined by Vector Copy Number
Time Frame: Up to 2 years
Reporting Status: Not Posted

7. Secondary Outcome: Identify Persistence of Transduced Myeloid Cells in Bone Marrow and Peripheral Blood as Determined by Vector Copy Number
Time Frame: At least 12 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Determine Clinical Response in Patients as Determined by IMWG Response Criteria
Time Frame: Up to 2 years
Reporting Status: Not Posted

9. Secondary Outcome: Fraction of Patients Achieving Complete Response With Minimal Residual Disease (MRD) Negativity
Time Frame: Up to 2 years
Reporting Status: Not Posted

10. Secondary Outcome: Determine Progression Free Survival in Patients
Time Frame: Up to 2 years
Reporting Status: Not Posted

11. Secondary Outcome: Determine Overall Survival in Patients
Time Frame: 2 years
Reporting Status: Not Posted

12. Secondary Outcome: Changes in Functional Status (Eastern Cooperative Oncology Group, ECOG)
Time Frame: 2 years
Reporting Status: Not Posted

13. Secondary Outcome: Changes in Functional Status (Karnofsky)
Time Frame: 2 years
Reporting Status: Not Posted

14. Secondary Outcome: Changes in Quality of Life: European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30
Time Frame: 2 years
Reporting Status: Not Posted

15. Secondary Outcome: Changes in Quality of Life: European Organisation for Research and Treatment of Cancer (EORTC) QLQ-MY20
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: No patients received Temferon
Description: No treatment related adverse events were reported as Temferon was not adminsitered
Groups:
- Untreated Patients: 3 patients recruited but did not receive Temferon
Arm/Group | Untreated Patients
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Although 3 patients were recruited, no patients received Temferon

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/95/NCT03875495/Prot_000.pdf